CLINICAL TRIAL: NCT06158347
Title: Efficacy and Safety of Hyperbaric Oxygen Therapy for Radiation Dermatitis in Patients with Localized Breast Cancer : a Randomized Controlled, Pilot Study
Brief Title: Efficacy and Safety of Hyperbaric Oxygen Therapy for Radiation Dermatitis in Patients with Localized Breast Cancer
Acronym: HBOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ilsan Cha hospital (Other)
Responsible Party: Principal Investigator, Jee Young Lee, assistant professor, CHA University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICICC-CT-23-01
Record Dates: First submitted 2023-11-06; First posted 2023-12-06 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Radiation Dermatitis
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HBOT group (Experimental): Hyperbaric oxygen therapy allows the patient to breathe 100% oxygen through an O2 Fresh M50 (HBOT Medical, Wonju, South Korea) chamber. Upon entering the chamber, oxygen is supplied while gradually increasing the atmospheric pressure from normal atmospheric pressure to 1.5 atmospheres absolute (ATA). If the intensity acceptable to the clinical research subject is lower than 1.5 ATA, maintain it at the point acceptable to the research subject and record that value.
  Interventions: Device: hyperbaric oxygen chamber
- control group (No Intervention): The control group will receive systemic education in dermal care and will be under the instruction of usual self-care.

INTERVENTIONS:
Device: hyperbaric oxygen chamber — Hyperbaric oxygen therapy allows patients to breathe 100% oxygen through an O2 Fresh M50 (HBOT Medical, Wonju, South Korea) chamber. Upon entering the chamber, oxygen is supplied by gradually increasing the barometric pressure from normal pressure to 1.5 atmospheres absolute (ATA).
  Arms: HBOT group

SUMMARY:
This study aimed to evaluate reducing the incidence of radiation dermatitis by assigning hyperbaric oxygen therapy to patients with localized breast cancer.

DETAILED DESCRIPTION:
To evaluate the efficacy of hyperbaric oxygen therapy (HBOT) on the prevention of radiation dermatitis, patients with localized breast cancer between the ages of 19 and 69 were randomly assigned to HBOT group and usual care group in a 1:1 ratio during the period of adjuvant radiotherapy.

The primary purpose of this study was to administer oxygen therapy three times a week during the radiotherapy period for those who were recommended to receive radiotherapy with a Biological equivalent dose (BED10) of 60 Gy or more as adjuvant radiotherapy after breast-conserving surgery to determine the radiation at the end of radiotherapy. The purpose is to compare the incidence of radiation dermatitis of therapy oncology group grade (RTOG grade) grade 2 or higher between the two groups.

The secondary purpose of this study is to evaluate/compare the following items in the relevant treatment group.

1. Comparison of the incidence of radiation dermatitis according to RTOG grade
2. Catterall skin scoring profile score comparison
3. Comparison of Skindex-29 questionnaire scores
4. Numeric rating scale score comparison
5. Investigation of radiation therapy dose, frequency, schedule, and medical history
6. Health-related quality of life questionnaire (EORTC-QLQ-C30)
7. Health-related quality of life measurement tool (EQ-5D)
8. Safety evaluation
9. Health-related quality of life measurement tool (EQ-5D)

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 19 and 69
2. Patients with biopsy confirmed invasive breast cancer
3. Patients who have undergone breast-conserving surgery for the purpose of tumor resection and require adjuvant radiotherapy or have undergone adjuvant radiotherapy within 5 times.
4. The Eastern Cooperative Oncology Group (ECOG) performance status 0-1
5. Those who understand the content of the study, agree to participate in the study, and provide written informed consent

Exclusion Criteria:

1. Subjects with distant metastases of cancer
2. Those whose cancer has invaded the skin of the breast (T4) or who have unhealed wounds on the skin
3. Patients who have a history of radiotherapy of the cervical thoracic region for other reasons in the past
4. Patients with a history of connective tissue disease
5. Subjects with uncontrolled diabetes with HbA1c 7.0 or higher
6. Pneumothorax and symptomatic upper respiratory tract infection
7. If it is judged that there will be a significant decrease in respiratory function
8. Undergoing treatments known to interact with hyperbaric oxygen therapy, such as cisplatin, doxorubicin, bleomycin, disulfiram, etc.
9. When it is judged that diseases other than cancer (dementia, cerebrovascular disease, severe renal failure, etc.) may have a significant effect on the decline of physical function.
10. If it is determined that the life expectancy is not sufficient follow-up within 3 months.
11. Pregnant and lactating women
12. Other persons who are judged by the researcher to be unsuitable for research

Ages: 19 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
incidence of grade 2 or more dermatitis according to RTOG toxicity scale | At the end of 6 weeks
  ① Grade 0: No change before or after treatment (No change over baseline)
  * Grade 1: Cystic lesions, erythema with faint or reduced skin luster, implantation, dry epidermis shedding, and decreased sweating.
  (Follicular, faint or dull erythema, epilation, dry desquamation, decreased sweating)
  * Grade 2: Tender or bright erythema, ecchymosis, desquamation of the wet epidermis, and moderate edema.
  (Tender or bright erythema, patchy moist desquamation, moderate edema)
  * Grade 3: Confluent skin lesions, desquamation of the wet epidermis other than the area where the skin is folded, pitting edema (Confluent, moist desquamation other than skin folds, pitting edema)
    * Grade 4: Ulcerative bleeding, skin necrosis (Ulceration hemorrhage, necrosis)

SECONDARY OUTCOMES:
RTOG toxicity | At the end of Day 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10
  ① Grade 0: No change before or after treatment (No change over baseline)
  * Grade 1: Cystic lesions, erythema with faint or reduced skin luster, implantation, dry epidermis shedding, and decreased sweating.
  (Follicular, faint or dull erythema, epilation, dry desquamation, decreased sweating)
  * Grade 2: Tender or bright erythema, ecchymosis, desquamation of the wet epidermis, and moderate edema.
  (Tender or bright erythema, patchy moist desquamation, moderate edema)
  * Grade 3: Confluent skin lesions, desquamation of the wet epidermis other than the area where the skin is folded, pitting edema (Confluent, moist desquamation other than skin folds, pitting edema)
    * Grade 4: Ulcerative bleeding, skin necrosis (Ulceration hemorrhage, necrosis)
CSSP | At the end of Day 1, week 5, week 8, week 9, week 10
  CSSP is a numerical scale-type evaluation tool developed by Fowler in 1965 to evaluate skin reactions in rats and modified by Catterall for application to patients with radiotherapy-induced dermatitis. [14] Graded from 1 to 10 points depending on the symptoms and severity of dermatitis
skindex-29 | At the end of Day 1, week 5, week 8, week 9, week 10
  Skindex-29 is a revision of the existing 61-item Skindex to 29 questions for patients with skin diseases. It maintains the excellent reproducibility, reliability, construct validity, and content validity of the Skindex, while improving the patient's quality of life through symptoms, function, and quality of life. It is a quality of life assessment tool designed to evaluate emotions on three scales. It consists of three scales: function (Fx), emotion (em), symptom (symptom) and a total score (total), linearly ranging from 0 (not affected) to 100 (always affected). A total of 29 items are scored for each scale, and then averaged to calculate the overall quality of life. The lower the score of Skindex-29, the better the quality of life.
NRS | At the end of Day 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10
  NRS is one of the evaluation tools that quantifies the level of discomfort. NRS 0 is defined as no discomfort, and NRS 10 is defined as the maximum discomfort the patient can think of.
EORTC | At the end of Day 1, week 5, week 8, week 9, week 10
  This is a questionnaire developed with 30 questions to measure the general quality of life of tumor patients. It evaluates overall quality of life and emotional health by dividing it into five areas: physical, role, cognitive, emotional, and social.
EQ-5D | At the end of Day 1, week 5, week 8, week 9, week 10
  It is the most widely used method of indirect measurement among various indirect measurement methods as it evaluates health status from multiple aspects, and then indirectly calculates the weight of the quality of a specific health status using a preference score assigned in advance for each functional level. The EQ-5D-5L consists of five questions, each of which asks about mobility, self-care, usual activities, pain, and anxiety/depression.
Drug Consumption | At the end of Day 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10
  The type, dose, route of administration, frequency, and purpose of medications administered or taken during the study period (medications prescribed due to current medical history or rescue drugs) will be recorded.
Adverse events | At the end of Day 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10
  To compare the occurrence of adverse events between the two groups and verify their safety. An adverse event is an undesirable or unintended sign, symptom, or disease that occurs after a procedure in a clinical study and does not necessarily have a causal relationship with the procedure. The investigator will analyze the incidence of adverse events, laboratory abnormalities, and serious adverse events that are suspected to be associated with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jee Youg Lee, Principal Investigator — Ilsan Cha hospital
Locations (1):
- Lee Jee Young, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JY, Hyun MH, Yang G, Lee S. Efficacy and safety of hyperbaric oxygen therapy for radiation-induced dermatitis in patients with breast cancer: a randomized pilot study. Support Care Cancer. 2025 Apr 21;33(5):399. doi: 10.1007/s00520-025-09463-0. PMID 40259026